CLINICAL TRIAL: NCT07095205
Title: Central Cholinergic Dysfunction in Depression: PET Imaging of a Novel Treatment Target With [18F]VAT to Assess the Antidepressant Effect of Nicotine
Brief Title: PET Imaging Using the Tracer [18F]VAT to Assess the Antidepressant Effect of Nicotine.
Acronym: VATMDDNicotine
Status: Recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Stony Brook University (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, Ramin Parsey, Professor of Psychiatry, Director of PET Strategy (M.D., Ph.D.), Stony Brook University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IRB2023-00490; 1R21MH137546-01 (NIH)
Record Dates: First submitted 2025-07-15; First posted 2025-07-31 (Actual); Last update posted 2025-07-31 (Actual); Status verified 2025-07

CONDITIONS: Major Depressive Disorder (MDD)
MeSH Terms: conditions — Depressive Disorder, Major | interventions — Tobacco Use Cessation Devices; Magnetic Resonance Spectroscopy

STUDY DESIGN:
Intervention Model Description: Participants diagnosed with Major Depressive Disorder (MDD) will receive two PET scans, one before and one after treatment. During the treatment period, participants with MDD will receive Nicorette NicoDerm CQ nicotine transdermal patches for 8 days (7 mg/day for days 1-2, 14 mg/day for days 3-4, and 21 mg/day for days 5-8). Non-depressed participants will have one PET scan and will not receive any nicotine treatment.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Control (Experimental): This arm consists of non-depressed participants. These participants will receive one PET scan utilizing tracer [18F] VAT to measure cholinergic terminal density.
  Interventions: Drug: PET Scan with [18F] VAT
- Major Depressive Disorder (MDD) (Experimental): This arm consists of participants diagnosed with Major Depressive Disorder. Participants in the MDD arm will receive interventional treatment for 8 days with transdermal nicotine patches. Participants in the MDD arm will also receive two PET scans with [18F]VAT tracer: one at baseline and one post-treatment.
  Interventions: Drug: Nicotine transdermal patch; Drug: PET Scan with [18F] VAT

INTERVENTIONS:
Drug: Nicotine transdermal patch — The participants with MDD will receive Nicorette NicoDerm CQ nicotine transdermal patches for 8 days (7 mg/day for days 1-2, 14 mg/day for days 3-4, and 21 mg/day for days 5-8).
  Other Names: Nicorette NicoDerm CQ; Nicotine patch
  Arms: Major Depressive Disorder (MDD)
Drug: PET Scan with [18F] VAT — All participants will undergo a PET scan at Baseline using tracer [18F] VAT. Participants with MDD will undergo a second post-treatment PET scan using tracer [18F] VAT.

SUMMARY:
In the brain, certain nerve cells communicate using a chemical called acetylcholine. Acetylcholine is thought to be important for several functions including mood, memory and wakefulness. The purpose of this study is to explore the role of these nerve cells in depression. Also, we would like to understand how nicotine, the study drug, works in depression and how it affects these nerve cells. To do this, brain imaging will be used before and after this treatment.

ELIGIBILITY:
Inclusion Criteria:

For Non-Depressed Participants:

* Age range 18 to 65 years old.
* Capacity to consent (able to read, understand, and sign informed consent).

For Participants with MDD

* Age range 18 to 65 years old.
* Capacity to consent (able to read, understand, and sign informed consent).
* Major Depressive Disorder (MDD) as primary diagnosis and currently in a major depressive episode
* Score of at least 29 on the Montgomery-Asberg Depression Rating Scale (MADRS).

Exclusion Criteria:

For Non-Depressed Participants:

* Nicotine use, including tobacco, e-cigarettes, nicotine patch, nicotine gum, within the past year [except for occasional users, who cannot use nicotine products in the week before the scan].
* Need for use of medication during the study that will affect cholinergic levels.
* Problematic drug/alcohol use that is judged sufficient to interfere with study procedures during the treatment period or impact participant safety.
* Significant active physical illness or neurological deficit that may affect brain function or imaging.
* Significant eye conditions such as keratoconus and/or need for rigid contact lenses.
* Current or lifetime history of a major psychiatric diagnosis.
* Any MRI contraindications, including recent tattoos, metal implants, pacemaker, metal prostheses, orthodontic appliances, or presence of shrapnel that are contraindicated for MRI.
* Any PET contraindications, including if study imaging will result in the participant receiving greater exposure than the research limit, or if participant is pregnant, currently breastfeeding, or planning to conceive during the course of study participation.
* Blood donation within 8 weeks of the [18F]VAT scan.

For Participants with MDD

* Nicotine use, including tobacco, e-cigarettes, nicotine patch, nicotine gum, within the past year [except for occasional users, who cannot use nicotine products in the week before the scan].
* Currently on effective antidepressant medications or need for use of medications that target the cholinergic system.
* Problematic drug/alcohol use that is judged sufficient to interfere with study procedures during the treatment period or impact participant safety.
* Significant active physical illness or neurological deficit that may affect the brain function or imaging.
* Significant eye conditions such as keratoconus and/or need for rigid contact lenses.
* Current or lifetime major psychiatric diagnosis other than MDD.
* Life-time history of psychosis or current psychosis.
* Significant risk for suicide.
* Any MRI contraindications, including recent tattoos, metal implants, pacemaker, metal prostheses, orthodontic appliances, or presence of shrapnel that are contraindicated for MRI.
* Any PET contraindications, including if study imaging will result in the participant receiving greater exposure than the research limit, or if participant is pregnant, currently breastfeeding, or planning to conceive during the course of study participation.
* Blood donation within 8 weeks of the [18F]VAT scan.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 14 (Estimated)
Dates: Start 2024-10-03 (Actual); Primary Completion 2029-09-30 (Estimated); Study Completion 2029-09-30 (Estimated)

PRIMARY OUTCOMES:
Change in Hamilton Depression Rating Scale-17 (HAMD) score. | Before and after 8 days of treatment with nicotine.
  Description: Comparison of Hamilton Depression Rating Scale-17 score at pretreatment and post-treatment. Minimum score 0, maximum possible score 52, with remission defined as <=7. The higher the score on the scale, the more severe the degree of depression.

CONTACTS AND LOCATIONS:
Overall Officials: Ramin Parsey, MD, PhD, Principal Investigator — Stony Brook University
Locations (1):
- Stony Brook University: Dept of Psychiatry, Stony Brook, New York, United States